CLINICAL TRIAL: NCT03107260
Title: The Association Between Variation in Oxygen Saturation (ScO2) and Incidence of Postoperative Cognitive Dysfunction (POCD) in a Population of Elderly Patients Admitted for Emergency Surgery.
Acronym: NIRS-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0018
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Cerebral Saturation; Cognitive Impairment; Emergencies
MeSH Terms: conditions — Cognitive Dysfunction; Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occurrence of postoperative cognitive dysfunction (Other)
  Interventions: Other: To evaluate the relationship between oxygen saturation and the incidence of postoperative cognitive dysfunction in emergency surgery in elderly patients

INTERVENTIONS:
Other: To evaluate the relationship between oxygen saturation and the incidence of postoperative cognitive dysfunction in emergency surgery in elderly patients — Evaluate the relationship between oxygen saturation and the incidence of postoperative cognitive dysfunction in non-cardiac, thoracic and vascular emergency surgery in patients 65 years of age and older. The occurrence of POCD will be defined by the MMSE decrease of at least 4 points at 24, 48 or 72 hours

SUMMARY:
There is no study of the association between ScO2 and POCD in non-cardiac, thoracic or vascular surgery. The few studies found in cardiac, thoracic and vascular surgery show an incidence up to 50% with a variation of the ScO2 threshold which varies between 15 and 25% according to the studies.

Age is the main risk of OCDD. The management of this pathology should be early to avoid loss of autonomy of the patient. Finding a relationship, if it exists, would therefore significantly improve the mortality and morbidity of the said patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Non-cardiac, thoracic and vascular emergency surgery
* Surgery under general anesthesia
* ASA I, II or III
* Simple information without consent
* Patient affiliated to social security

Exclusion Criteria:

* Inability to understand
* Patient under tutelage, or curatorship or deprived of public right
* ASA IV
* History of severe dementia MMSE <20
* Personal or familial history of malignant hyperthermia
* History of allergy or hypersensitivity to anesthetic products used
* Contra-indication to Cisatracurium®: myasthenia gravis
* Contra-indication to Sevoflurane®
* Contra-indication to local anesthetics
* Indication of use of a Ketamine®-type hypnotic (modification of the BIS)
* Indication of use of nitrous oxide
* History of cranial trauma
* Neuromuscular pathology
* Spinal anesthesia
* Cardiac, thoracic or vascular surgery
* Surgery not performed in emergency
* Neurochirugia in the context of cranial trauma
* Any surgery that does not allow the use of the NIRS (impossibility of positioning of the electrodes by the location of the surgical field).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-01-15 (Actual); Primary Completion 2018-07-13 (Estimated); Study Completion 2018-07-13 (Estimated)

PRIMARY OUTCOMES:
Occurrence of POCD | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France